CLINICAL TRIAL: NCT01995669
Title: A Phase I/II Study of Lenalidomide and Obinutuzumab (GA101) in Relapsed Indolent Non-Hodgkin's Lymphoma
Brief Title: Lenalidomide and Obinutuzumab in Treating Patients With Relapsed Indolent Non-Hodgkin Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-0261; NCI-2014-00943 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ML28301; 2013-0261 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2013-11-20; First posted 2013-11-26 (Estimated); Results first posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Grade 3a Follicular Lymphoma; Recurrent Follicular Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Small Lymphocytic Lymphoma; Refractory Follicular Lymphoma; Refractory Marginal Zone Lymphoma; Refractory Small Lymphocytic Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Lenalidomide; obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (lenalidomide, obinutuzumab) (Experimental): Patients receive lenalidomide PO QD on days on days 2-22 and obinutuzumab IV over 4-5 hours on days 1, 2, 8, 15, and 22 of cycle 1 and on day 1 of each subsequent cycle. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients not experiencing progression and who in the opinion of treating physician are deriving benefit from combination treatment may continue lenalidomide for an additional 6 cycles (up to cycle 12) and obinutuzumab on day 1 every 2 months for up to 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Lenalidomide; Biological: Obinutuzumab

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Lenalidomide — Given PO
  Other Names: CC-5013; CC5013; CDC 501; Revlimid
Biological: Obinutuzumab — Given IV
  Other Names: Anti-CD20 Monoclonal Antibody R7159; GA-101; GA101; Gazyva; huMAB(CD20); R7159; RO 5072759; RO-5072759; RO5072759

SUMMARY:
This phase I/II trial studies the side effects and best dose of lenalidomide when given together with obinutuzumab and how well this combination works in treating patients with low-grade non-Hodgkin lymphoma (NHL) that has returned after a period of improvement (relapsed). Biological therapies, such as lenalidomide, may attack specific cancer cells and stop them from growing or kill them. Obinutuzumab is a form of targeted therapy because it attaches itself to specific molecules (receptors) on the surface of cancer cells, known as CD20 receptors. When obinutuzumab attaches to CD20 receptors, the signals that tell the cells to grow are blocked and the cancer cell may be marked for destruction by the body's immune system. Giving lenalidomide and obinutuzumab together may work better in treating NHL.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose of lenalidomide plus obinutuzumab in relapsed/refractory indolent lymphoma. (Phase I) II. To evaluate the safety of lenalidomide in combination with obinutuzumab in patients with relapsed/refractory indolent lymphoma. (Phase II) III. To determine the overall response rate (ORR) of the combination in patients with relapsed/refractory indolent lymphoma. (Phase II)

SECONDARY OBJECTIVES:

I. To determine the complete response rate, time to progression (TTP), and progression free survival in patients with indolent lymphoma following treatment with obinutuzumab + lenalidomide.

II. To evaluate changes in immune effector cells and the tumor microenvironment following treatment with obinutuzumab + lenalidomide.

OUTLINE: This is a phase I, dose-escalation study of lenalidomide followed by a phase II study.

Patients receive lenalidomide orally (PO) once daily (QD) on days 2-22 and obinutuzumab intravenously (IV) over 4-5 hours on days 1, 2, 8, 15, and 22 of cycle 1 and on day 1 of each subsequent cycle. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients not experiencing progression and who in the opinion of treating physician are deriving benefit from combination treatment may continue lenalidomide for an additional 6 cycles (up to cycle 12) and obinutuzumab on day 1 every 2 months for up to 2 years in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 1 year, every 6 months for 1 year, and then yearly thereafter.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of small lymphocytic lymphoma, follicular lymphoma (grades 1-3a), or marginal zone lymphoma
* Evidence of progression or lack of response following at least 1 prior treatment for indolent lymphoma
* Able and willing to provide written informed consent and to comply with the study protocol
* Must have at least 1 node greater than 1.5 cm in short axis diameter
* Adequate hematologic function (unless abnormalities are related to NHL), defined as follows:
* Hemoglobin >= 9.0 g/dL
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L; ANC < 1.5 x 10^9/L if cytopenia is due to extensive bone marrow involvement of disease as determined by the treating physician
* Platelet count (PLT) >= 75 x 10^9/L; PLT count less than 100 x 10^9/L if cytopenia is due to extensive bone marrow involvement of disease as determined by the treating physician
* For men who are not surgically sterile, agreement to use a barrier method of contraception for >= 3 months after the last obinutuzumab dose; in addition, male patients must agree to request that their partners use an additional method of contraception, such as oral contraceptives, intrauterine device, barrier method of contraception, or spermicidal jelly
* For women of reproductive potential who are not surgically sterile, agreement to use two adequate methods of contraception, such as oral contraceptives, intrauterine device, or barrier method of contraception in conjunction with spermicidal jelly for >= 12 months after the last obinutuzumab dose
* Females of childbearing potential (FCBP) must have a negative serum pregnancy test with a sensitivity of at least 50 mIU/mL within 10-14 days prior to and again within 24 hours of prescribing lenalidomide and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 4 weeks before she starts taking lenalidomide; FCBP must also agree to ongoing pregnancy testing; men must agree to use a latex condom during sexual contact with a female of child bearing potential even if they have had a successful vasectomy

  * A female of childbearing potential is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
* All study participants must be registered into the mandatory Revlimid Risk Evaluation and Mitigation Strategy (REMS) program, and be willing and able to comply with the requirements of Revlimid REMS program
* For patients with bulky disease (tumors > 5 cm); must be able to take aspirin (81 mg or 325 mg) daily as prophylactic anticoagulation (patients intolerant to acetylsalicylic acid [ASA] may use warfarin or low molecular weight heparin)
* Females of reproductive potential must adhere to the scheduled pregnancy testing as required in the Revlimid REMS program; able to take aspirin (81 or 325 mg) daily as prophylactic anticoagulation (patients intolerant to ASA may use warfarin or low molecular weight heparin)

Exclusion Criteria:

* Evidence ongoing transformation into aggressive NHL
* History of severe allergic or anaphylactic reactions to monoclonal antibody therapy
* Known hypersensitivity to thalidomide or lenalidomide
* Regular treatment with corticosteroids during the 4 weeks prior to the start of cycle 1, unless administered for indications other than NHL at a dose equivalent to =< 30 mg/day prednisone
* History of prior malignancy within the last 5 years, with the exception of curatively treated basal or squamous cell carcinoma of the skin and low-grade in situ carcinoma of the cervix
* Evidence or history of significant, uncontrolled concomitant diseases that could affect compliance with the protocol or interpretation of results, including significant cardiovascular disease (such as New York Heart Association class III or IV cardiac disease, severe arrhythmia, myocardial infarction within the previous 6 months, unstable arrhythmias, or unstable angina) or pulmonary disease (including obstructive pulmonary disease and history of bronchospasm)
* Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds) or any major episode of infection requiring treatment with IV antibiotics or hospitalization (relating to the completion of the course of antibiotics, except if for tumor fever) within 4 weeks prior to the start of cycle 1; patients with suspected active or latent tuberculosis (latent tuberculosis needs to be confirmed by positive interferon-gamma release assay)
* Vaccination with live vaccines within 28 days prior to start of treatment
* Any of the following abnormal laboratory values (unless any of these abnormalities are due to underlying lymphoma)
* Creatinine > 1.5 times the upper limit of normal (ULN) (unless creatinine clearance normal), or calculated creatinine clearance < 40 mL/min (using Cockcroft-Gault formula)
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2.5 x ULN
* Total bilirubin > 1.5 x ULN (or > 3 x ULN for patients with documented Gilbert syndrome)
* Any history of hepatitis B infection
* Positive test results for hepatitis C (hepatitis C virus [HCV] antibody serology testing); patients positive for HCV antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV ribonucleic acid (RNA)
* Known history of human immunodeficiency virus (HIV) seropositive status
* Positive test results for human T-lymphotropic 1 (HTLV 1) virus; HTLV testing is required in patients from endemic countries (Japan, countries in the Caribbean basin, South America, Central America, Sub Saharan Africa, and Melanesia)
* Pregnant or lactating
* Eastern Cooperative Oncology Group (ECOG) performance status greater than 2
* Participation in another clinical trial with drug intervention within 21 days prior to start of cycle 1 and during the study
* Patients with small lymphocytic lymphoma (SLL)/chronic lymphocytic leukemia (CLL) are excluded during the phase I portion of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2014-05-27 (Actual); Primary Completion 2023-01-23 (Actual); Study Completion 2023-01-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Loretta Nastoupil, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Gurumurthi A, Chin CK, Feng L, Fowler NH, Strati P, Hagemeister FB, Fayad LE, Westin JR, Obi C, Arafat J, Nair R, Steiner RE, Neelapu SS, Flowers CR, Nastoupil LJ. Safety and activity of lenalidomide in combination with obinutuzumab in patients with relapsed indolent non-Hodgkin lymphoma: a single group, open-label, phase 1/2 trial. EClinicalMedicine. 2024 Jul 27;74:102747. doi: 10.1016/j.eclinm.2024.102747. eCollection 2024 Aug. PMID 39161543
- See also: University of Texas MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled into an investigator initiated, open-label, phase 1/2 trial at a single institution, MD Anderson Cancer Center, Houston, TX, US.
Groups:
- Phase I Dose Level 10mg Lenolidomide + 1000mg Obinutuzimab: Participants with relapsed or refractory WHO Grade 1 to 3A follicular lymphoma
- Phase I Dose Level 15mg Lenolidomide + 1000mg Obinutuzimab; Phase I Dose Level 20mg Lenolidomide + 1000mg Obinutuzimab: Patients with relapsed or refractory WHO Grade 1 to 3A follicular lymphoma
- Phase II: Expansion Len 20 mg Plus Obin 1000 mg: Participants with relapsed or refractory WHO Grade 1 to 3A follicular lymphoma, marginal zone lymphoma and small lymphocytic lymphoma
Period: Overall Study
Arm/Group | Phase I Dose Level 10mg Lenolidomide + 1000mg Obinutuzimab | Phase I Dose Level 15mg Lenolidomide + 1000mg Obinutuzimab | Phase I Dose Level 20mg Lenolidomide + 1000mg Obinutuzimab | Phase II: Expansion Len 20 mg Plus Obin 1000 mg
Started | 3 | 3 | 3 | 57
Completed | 1 | 2 | 2 | 28
Not Completed | 2 | 1 | 1 | 29
Not completed — Progression | 2 | 1 | 1 | 13
Not completed — Adverse Event | 0 | 0 | 0 | 3
Not completed — Death | 0 | 0 | 0 | 6
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 6
Not completed — Insurance Expired | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Phase I Dose Level 10mg Lenolidomide + 1000mg Obinutuzimab; Phase I Dose Level 15mg Lenolidomide + 1000mg Obinutuzimab; Phase I Dose Level 20mg Lenolidomide + 1000mg Obinutuzimab: Patients with relapsed or refractory WHO Grade 1 to 3A follicular lymphoma
- Ph. II: Expansion Len 20 mg Plus Obin 1000 mg: Participants with relapsed or refractory WHO Grade 1 to 3A follicular lymphoma, marginal zone lymphoma and small lymphocytic lymphoma
- Total: Total of all reporting groups
Arm/Group | Phase I Dose Level 10mg Lenolidomide + 1000mg Obinutuzimab | Phase I Dose Level 15mg Lenolidomide + 1000mg Obinutuzimab | Phase I Dose Level 20mg Lenolidomide + 1000mg Obinutuzimab | Ph. II: Expansion Len 20 mg Plus Obin 1000 mg | Total
Number analyzed (Participants) | 3 | 3 | 3 | 57 | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 1 | 0 | 32 | 36
  >=65 years | 0 | 2 | 3 | 25 | 30
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1 | 28 | 30
  Male | 2 | 3 | 2 | 29 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 7 | 7
  Not Hispanic or Latino | 3 | 3 | 3 | 50 | 59
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 3 | 4
  White | 2 | 3 | 2 | 54 | 61
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 3 | 3 | 57 | 66

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose of Lenalidomide When Given With Obinutuzumab Defined as the Highest Dose Level Have Been Treated With Less Than 2 Instances of Dose Limiting Toxicity DLT.
Description: To determine the maximum tolerated dose of lenalidomide plus obinutuzumab in relapsed/refractory indolent lymphoma the 3 by 3 method was used. (Phase I) Doses of Lenalidomide to be used are 10mg, 15mg, 20mg in Phase 1.
Time Frame: 28 days after 168 days (6 courses)
Population: Phase II was not assessed.
Measure: Number; unit: mg
Groups:
- All Participants: Phase I Dose Level 10mg Lenolidomide + 1000mg Obinutuzimab Phase I Dose Level 15mg Lenolidomide + 1000mg Obinutuzimab Phase I Dose Level 20mg Lenolidomide + 1000mg Obinutuzimab
Arm/Group | All Participants
Number analyzed (Participants) | 9
mg | 20

2. Secondary Outcome: Overall Survival, Time to Progression, and Progression Free Survival (Phase II)
Description: The distribution of time-to-event endpoints will be estimated using the method of Kaplan and Meier. Comparison of time-to-event endpoints by important subgroups will be made using the log-rank test.The distribution of time-to-event endpoints will be estimated using the method of Kaplan and Meier. Comparison of time-to-event endpoints by important subgroups will be made using the log-rank test.
Time Frame: up to 4 years
Population: Phase I was not assessed for this outcome.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ph. II: Expansion Len 20 mg Plus Obin 1000 mg
Number analyzed (Participants) | 57
months
  PFS | 44.2 [22.5 to NA] — Median PFS was not reached due to insufficient number of patients with events.
  OS | NA [NA to NA] — Median OS was not reached due to insufficient number of patients with events.
  TTP | 44.2 [26.6 to NA] — Median TTP was not reached due to insufficient number of patients with events.

ADVERSE EVENTS:
Time Frame: from consent up to 30 days post last dose, up to 4 years
Arm/Group | Phase I Dose Level 10mg Lenolidomide + 1000mg Obinutuzimab | Phase I Dose Level 15mg Lenolidomide + 1000mg Obinutuzimab | Phase I Dose Level 20mg Lenolidomide + 1000mg Obinutuzimab | Ph. II: Expansion Len 20 mg Plus Obin 1000 mg
All-Cause Mortality (participants affected / at risk) | 0/3 | 1/3 | 0/3 | 6/57
Serious Adverse Events (participants affected / at risk) | 1/3 | 3/3 | 1/3 | 34/57
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 57/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I Dose Level 10mg Lenolidomide + 1000mg Obinutuzimab (N=3) | Phase I Dose Level 15mg Lenolidomide + 1000mg Obinutuzimab (N=3) | Phase I Dose Level 20mg Lenolidomide + 1000mg Obinutuzimab (N=3) | Ph. II: Expansion Len 20 mg Plus Obin 1000 mg (N=57)
Lung Infection (Infections and infestations) | 1 (1) | 0 | 0 | 5 (8)
Sepsis (Infections and infestations) | 0 | 3 (3) | 0 | 3 (3)
Appendicitis (Infections and infestations) | 0 | 1 (1) | 0 | 1
Unintented Pregnancy (Reproductive system and breast disorders) | 0 | 1 (1) | 0 | 0
Gastroeophogeal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 0
Hyperglycemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 (1)
Tumor Lysis Syndrome (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1
Chest pain (Cardiac disorders) | 0 | 0 | 1 | 1 (1)
Hypotension (Cardiac disorders) | 0 | 0 | 0 | 1
Sick Sinus Syndrome (Cardiac disorders) | 0 | 0 | 0 | 1
Sinus Tackycardia (Cardiac disorders) | 0 | 0 | 0 | 2 (2)
Syncope (Cardiac disorders) | 0 | 0 | 0 | 1 (1)
Fever (General disorders) | 0 | 0 | 0 | 1 (2)
Heart Faliure (General disorders) | 0 | 0 | 0 | 1 (1)
Pacemaker implant (General disorders) | 0 | 0 | 0 | 2 (2)
Bactermia (Infections and infestations) | 0 | 0 | 0 | 1 (1)
Cellulitis - left Mandible (Infections and infestations) | 0 | 0 | 0 | 1 (1)
Cellulitis - right calf (Infections and infestations) | 0 | 0 | 0 | 1 (1)
Infection - JC Virus (Infections and infestations) | 0 | 0 | 0 | 1 (1)
Infection, pacemaker infection (Infections and infestations) | 0 | 0 | 0 | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 (1)
Gait disturbance (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 (1)
Vertigo (Nervous system disorders) | 0 | 0 | 0 | 1 (1)
Gallbladder obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 1 (1)
Reproductive system and breast disorder - testicular pain and dysuria (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 (1)
Squamous Cell Carcinoma (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I Dose Level 10mg Lenolidomide + 1000mg Obinutuzimab (N=3) | Phase I Dose Level 15mg Lenolidomide + 1000mg Obinutuzimab (N=3) | Phase I Dose Level 20mg Lenolidomide + 1000mg Obinutuzimab (N=3) | Ph. II: Expansion Len 20 mg Plus Obin 1000 mg (N=57)
Abdominal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (6)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Allergic reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 8 (8)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0) | 11 (12)
Anxiety (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Appetite Change, Increase (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 14 (19)
Bloating (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Blurred Vision (General disorders) | 1 (1) | 1 (2) | 1 (1) | 12 (13)
Cataract (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Chills (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 5 (5)
Confusion (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (2) | 2 (6) | 25 (44)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 1 (2) | 33 (48)
Creatinine increased (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deconditioning (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased Visual Acuity (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (9) | 2 (7) | 2 (7) | 23 (55)
Dizziness (General disorders) | 3 (5) | 0 (0) | 1 (1) | 19 (29)
Dry Eye (Eye disorders) | 2 (2) | 0 (0) | 1 (1) | 15 (19)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 3 (4) | 2 (10) | 18 (27)
Edema - Face (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 6 (10)
Edema - Limbs (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 22 (30)
Edema - Trunk (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 4 (5)
Eye disorders - Double Vision (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Eye disorders -Watery eye (1 #9) (General disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Eye Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Eye Stye (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Fatigue (General disorders) | 3 (21) | 2 (13) | 2 (8) | 50 (112)
Fever (General disorders) | 1 (1) | 0 (0) | 0 (0) | 16 (26)
Flatulence (Gastrointestinal disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Floaters (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flu-like symptoms (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flushing (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Gallbladder obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Glaucoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (General disorders) | 1 (1) | 1 (1) | 0 (0) | 8 (11)
Heart Failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic enzyme elevation (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypogammaglobulinemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0) | 3 (3)
Hypokalemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypertension (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypomagnesmia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Indigestion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Infections and infestations - Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Investigations Other - Elevated LDH (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 5 (8)
Lymphocyte count decreased (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Memory Impairment (General disorders) | 1 (2) | 1 (1) | 2 (4) | 11 (16)
Mucositis Oral (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 11 (15)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1) | 2 (12) | 25 (49)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (5) | 1 (2) | 20 (30)
Neutrophil Count Decreased (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 15 (33)
Oral Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pacemaker Placed (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 16 (20)
Platelet count decreased (Blood and lymphatic system disorders) | 2 (2) | 2 (3) | 1 (1) | 11 (21)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (4) | 8 (9)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 35 (60)
Respiratory, thoracic and mediastinal disorders - Chest congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 11 (12)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Sinus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 10 (13)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thromboembolic event (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tinnitus (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 2 (3) | 2 (2)
Twitching (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Unintended Pregnancy (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 8 (10)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
White Blood Cell Decreased (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (4)
Hearing Impaired (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hot flashes (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypersensitive smell (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Localized edema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paresthesia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sleep disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Swollen eye (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toothache (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Visual disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Watering eyes (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Weight gain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight loss (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Migraine (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bacteremia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Facial Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mycobacterial Avium infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 9 (10)
Epididymoorchitis with possible abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Scratchy throat-closing (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Shingles (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Staph infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gait disturbance (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (8)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (7)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Testicular pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Right toe strain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Difficulty Urinating (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Polyuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal Insufficiency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Urinary urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaginal discharge (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal cell carcinoma (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythroderma (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insect bite (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Skin infection (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Squamous cell carcinoma (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Wasp bite (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abcess (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Color change on abdomen (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Plantar's wart (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Plaque psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-11): https://cdn.clinicaltrials.gov/large-docs/69/NCT01995669/Prot_SAP_000.pdf